CLINICAL TRIAL: NCT04356937
Title: Tocilizumab to Prevent the Progression of Hypoxemic Respiratory Failure in Hospitalized Non-Critically Ill Patients With COVID-19
Brief Title: Efficacy of Tocilizumab on Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Stone, John H, M.D., M.P.H, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P001159
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: SARS-CoV 2
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized,double blind, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Subjects who meet all inclusion criteria and none of the exclusion criteria will be randomized 2:1 to tocilizumab or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (Experimental): Review effect of Tocilizumab on multi-organ dysfunction in a phase 3 randomized controlled trial among hospitalized patients with COVID-19 infection.
  Participants will receive an intravenous (IV) injection of 8 mg/kg (not to exceed 800 mg) tocilizumab.Specifically, as compared to placebo, we will test whether tocilizumab is associated with a reduction in multi-organ dysfunction among hospitalized COVID-19 adult patients with elevated inflammatory measures.
  Interventions: Drug: Tocilizumab
- Standard of care plus placebo (Placebo Comparator): Participants will receive an placebo intravenous (IV) injection of 8 mg/kg (not to exceed 800 mg).Specifically, as compared to placebo, we will test whether tocilizumab is associated with a reduction in multi-organ dysfunction among hospitalized COVID-19 adult patients with elevated inflammatory measures.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tocilizumab — Patients will receive the standard treatment for COVID-19 per MGH guidance and also be randomized (2:1) to one of the following arms:
  1. Tocilizumab 8mg x 1 (n=185)
  2. Standard of care/Placebo (n=93)
  Other Names: Actemra
  Arms: Tocilizumab
Drug: Placebos — Patients will receive the standard treatment for COVID-19 per MGH guidance and also be randomized (2:1) to one of the following arms:
  1. Tocilizumab 8mg x 1 (n=185)
  2. Standard of care/Placebo (n=93)
  Arms: Standard of care plus placebo

SUMMARY:
This is a randomized, double blind, multi-center study to evaluate the effects of tocilizumab compared to placebo on patient outcomes in participants with confirmed SARS-CoV-2 infection and evidence of systemic inflammation.

The aim of this study is to test the effect of Tocilizumab on multi-organ dysfunction in a phase 3 randomized controlled trial among hospitalized patients with COVID-19 infection.

Specifically, as compared to placebo, we will test whether tocilizumab is associated with a reduction in multi-organ dysfunction among hospitalized COVID-19 adult patients with elevated inflammatory measures. Multi-organ dysfunction will be measured as the incidence of the following composite endpoint (mechanical ventilation, renal replacement therapy, mechanical support, need for inotropes or vasopressors, liver dysfunction (increased bilirubin), and all-cause mortality). We will also assess multiple pre-specified secondary (exploratory) endpoints and safety endpoints.

We hypothesize that, as compared to placebo, tocilizumab will reduce transfer to the ICU, need for mechanical ventilation, increase rates of hospital discharge in patients diagnosed with severe COVID-19 infection and evidence of exaggerated inflammatory response.

DETAILED DESCRIPTION:
As of April 3, 2020, COVID-19 has been confirmed in over 1 million people worldwide, with an estimated symptomatic case fatality ratio of around 1.4%. Currently without an effective treatment for SARS-CoV-2 there is an urgent need for effective treatment to curtail the rate of respiratory failure, the leading cause of mortality in COVID-19 disease. Moreover, with increasing numbers of patients requiring intensive unit level care and mechanical ventilation, nations are already having to triage patients for ventilatory support due to limited resources and healthcare systems around the world being stretched to the point of collapse, highlighting the importance of identifying interventions that could prevent the development of respiratory failure for these patients.

The disease course of COVID-19 includes an incubation period, an acute viral phase that most commonly presents with flu-like symptoms that in some individuals progresses to a severe hyperinflammatory phase marked by acute respiratory distress syndrome (ARDS) and hypoxemic respiratory failure.Though there is spectrum of clinical course, many progress to the hyperinflammatory phase around day seven of symptoms, often requiring intensive care unit (ICU) level care and mechanical ventilation. Accumulating evidence suggests that the pathophysiology underlying this profound decline is a severe inflammatory response as demonstrated by multi organ system dysfunction akin to cytokine release syndrome (CRS)/macrophage activation syndrome (MAS).CRS/MAS is a systemic hyperinflammatory syndrome on a spectrum with secondary hemophagocytic lymphohistiocytosis (sHLH), typically characterized by multiorgan failure that is often triggered by viral infections in the setting of excessive immune activation, typically with marked hyperferritinemia.Postmortem assessment of patients with COVID-19 have demonstrated pathologic findings consistent with MAS such as mono/lymphocytic infiltrates within the lung parenchyma with associated edema and alveolar congestion, splenic necrosis with macrophage proliferation and hemophagocytosis, as well as a lymphocyte/histiocyte predominate infiltrate of portal vasculature accompanying liver necrosis and sinusoidal congestion.Cytokine profiling of patients with MAS/sHLH overlaps with that seen in patients with severe COVID-19 and includes elevated levels of IL-1, IL-2, IL-7, IL-6, G-CSF, MCP- 1, and TNF-α as well as elevated D-dimer, C-reactive protein, LDH and troponins.Moreover, preliminary data from a non-randomized series of COVID-19 patients with "severe or critical COVID-19" from China who were treated with tocilizumab (in addition to standard therapies) showed they had dramatic improvement in fever, arterial oxygen saturation and inflammatory markers within the first 24-hours following administration.

Taken together, these data strongly suggest an immunologic link between COVID-19 and immune dysregulation resulting in MAS. Clinical trials are already underway studying the role of immunomodulatory therapy including modulation of IL-1 and IL-6 and downstream pathways in the setting of CAR-T induced MAS (NCT04150913, NCT04071366) and agents such anakinra and tocilizumab have been used in this context with promising results and good safety profiles. There is an urgent and dire need to study the therapeutic role for immunomodulatory therapy in COVID-19 disease to both halt disease progression in patients at an individual level and prevent the inevitable saturation of healthcare resources at a systems level, to which end there are numerous ongoing international trials to expand these efforts into the setting of COVID-19 infection (ChiCTR2000029765, NCT04324021, TOCOVID-19). Based on the MGH experience thus far with COVID-19, including over 200 patients to date, the need for mechanical ventilation has been approximately 30%. With the upcoming surge anticipated between April 17th and 21st we expect the need for hundreds of additional ICU beds. Investigators propose a trial of IL-6 receptor blockade with tocilizumab given early in disease course to try to prevent progression of COVID-19.

ELIGIBILITY:
Inclusion criteria:

Subjects who meet all of the following criteria will be eligible to participate in the study:

1. Must have provided informed consent in a manner approved by the Investigator's Institutional Review Board (IRB) or Independent Ethics Committee (IEC) prior to any assessments. If a patient is unable to provide informed consent due to their medical condition, the patient's legally authorized representative may consent on behalf of the study patient, as permitted by local law and institutional Standard Operating Procedures;
2. Age Range: 19-85 years old
3. Male or female gender
4. Confirmed SARS-CoV-2 infection by nasopharyngeal swab PCR or serum assay for IgM antibody
5. Requiring hospital but not mechanical ventilation
6. Oxygen supplementation not greater than 10L delivered by any device
7. WITH evidence of severe COVID-19 (at least 2 of the following):

   1. Fever > 38C within 72 hours
   2. Pulmonary infiltrate on CXR
   3. Need for supplemental O2 to maintain saturation > 92%
8. AND at least 1 of the following:

   1. Ferritin > 500 ng/ml
   2. CRP > 50 mg/L
   3. LDH >250 U/L
   4. D-dimer > 1000 ng/mL
9. Women of childbearing potential (ie, not post-menopausal or surgically sterilized) must have a negative highly sensitive urine or serum pregnancy test before randomization. Participating women of childbearing potential must be willing to consistently use effective methods of contraception (ie, condom, combined oral contraceptive, implant, injectable, indwelling intrauterine device, or a vasectomized partner) from screening until at least 90 days after administration of the last dose of study drug;
10. The subject must be willing and able to provide informed consent and abide all study requirements and restrictions.

Exclusion criteria:

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Unable to provide verbal informed consent or have verbal agreement to participate through attestation and signature of a Witness required, as outlined in the Partners IRB's Table for Consenting in COVID Research that is More than Minimal Risk.
2. Subjects between the ages of 79 and 86 will be excluded if they have NYHA Class III/IV heart failure, insulin-dependent diabetes mellitus, angina, or treatment of a malignancy (excluding non-melanoma skin cancer) within six months
3. Uncontrolled bacterial, fungal, or non-COVID viral infection
4. Active TB
5. Any prior investigational immunosuppressive therapy within 28-days or 3 half-lives of the agent (for instance with biologic or JAK inhibitor)
6. Any concurrent immunosuppressive medication that the PI believes would put the patient at higher risk
7. Receipt of intravenous tocilizumab for the treatment of a non-COVID condition within three weeks of the first COVID symptom
8. History of hypersensitivity to tocilizumab
9. Any concurrent immunosuppressive medication that the PI believes would put the patient at higher risk
10. Treatment with other biologic or small-molecule immunosuppressive therapy such as IL1R-antagonism, JAK inhibition, or other agents
11. Treatment with convalescent plasma
12. History of diverticulitis or bowel perforation
13. ANC <500, Platelets <50,000*
14. AST/ALT > 5X ULN
15. Women who are pregnant or planning to get pregnant in the next 90 days;
16. Any condition that could interfere with, or for Known allergy to the study drug or any of its ingredients or known allergy to any other anti IL 6 agents;
17. Any condition that could interfere with or for which the treatment might interfere with, the conduct of the study or interpretation of the study results, or that would, in the opinion of the Investigator, increase the risk of the subject by participating in the study.

We note that anti-viral therapies may be administered to subjects if given in the context of a clinical trial. Nitric oxide treatment is also permitted at the discretion of the care team, ideally in the context of a clinical trial. Co-treatment chloroquine, hydroxychloroquine, and/or azithromycin is permitted for subjects in this protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Stone, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Request for IPD can be submitted to PI for review

REFERENCES:
- [Derived] Stone JH, Frigault MJ, Serling-Boyd NJ, Fernandes AD, Harvey L, Foulkes AS, Horick NK, Healy BC, Shah R, Bensaci AM, Woolley AE, Nikiforow S, Lin N, Sagar M, Schrager H, Huckins DS, Axelrod M, Pincus MD, Fleisher J, Sacks CA, Dougan M, North CM, Halvorsen YD, Thurber TK, Dagher Z, Scherer A, Wallwork RS, Kim AY, Schoenfeld S, Sen P, Neilan TG, Perugino CA, Unizony SH, Collier DS, Matza MA, Yinh JM, Bowman KA, Meyerowitz E, Zafar A, Drobni ZD, Bolster MB, Kohler M, D'Silva KM, Dau J, Lockwood MM, Cubbison C, Weber BN, Mansour MK; BACC Bay Tocilizumab Trial Investigators. Efficacy of Tocilizumab in Patients Hospitalized with Covid-19. N Engl J Med. 2020 Dec 10;383(24):2333-2344. doi: 10.1056/NEJMoa2028836. Epub 2020 Oct 21. PMID 33085857

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Standard care plus a single dose of tocilizumab (8 mg/kg administered intravenously, not to exceed 800 mg)
- Placebo: Standard care plus placebo
Period: Randomization (Safety Population)
Arm/Group | Tocilizumab | Placebo
Started | 161 | 82
Completed | 161 | 82
Not Completed | 0 | 0
Period: Treatment (mITT Population)
Arm/Group | Tocilizumab | Placebo
Started | 161 | 82
Completed | 161 | 81
Not Completed | 0 | 1
Not completed — Intubated before receiving study treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Tocilizumab: Review effect of Tocilizumab on multi-organ dysfunction in a phase 3 randomized controlled trial among hospitalized patients with COVID-19 infection.
  Participants will receive an intravenous (IV) injection of 8 mg/kg (not to exceed 800 mg) tocilizumab. Specifically, as compared to placebo, we will test whether tocilizumab is associated with a reduction in multi-organ dysfunction among hospitalized COVID-19 adult patients with elevated inflammatory measures.
  Tocilizumab: Patients will receive the standard treatment for COVID-19 per MGH guidance and also be randomized (2:1) to one of the following arms:
  1. Tocilizumab 8mg x 1
  2. Standard of care/Placebo
- Standard of Care Plus Placebo: Participants will receive an placebo intravenous (IV) injection of 8 mg/kg (not to exceed 800 mg).Specifically, as compared to placebo, we will test whether tocilizumab is associated with a reduction in multi-organ dysfunction among hospitalized COVID-19 adult patients with elevated inflammatory measures.
  Placebos: Patients will receive the standard treatment for COVID-19 per MGH guidance and also be randomized (2:1) to one of the following arms:
  1. Tocilizumab 8mg x 1
  2. Standard of care/Placebo
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Standard of Care Plus Placebo | Total
Number analyzed (Participants) | 161 | 82 | 243
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.6 [46.4 to 69.7] | 56.5 [44.7 to 67.8] | 59.8 [45.3 to 69.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 37 | 102
  Male | 96 | 45 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 39 | 109
  Not Hispanic or Latino | 84 | 35 | 119
  Unknown or Not Reported | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or ethnic group: American Indian or Alaska Native | 1 | 0 | 1
  Race or ethnic group: Asian | 7 | 2 | 9
  Race or ethnic group: Black | 24 | 16 | 40
  Race or ethnic group: Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Race or ethnic group: White | 71 | 33 | 104
  Race or ethnic group: Other | 35 | 15 | 50
  Race or ethnic group: Unknown | 23 | 15 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161 | 82 | 243
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.9 [26.0 to 34.2] | 30.2 [25.7 to 33.8] | 30.1 [25.9 to 34.2]
BMI ≥ 30 kg/m^2 [Count of Participants; unit: Participants] | 80 | 42 | 122
Days from symptom onset to randomization [Median (Inter-Quartile Range); unit: days] | 9.0 [6.0 to 13.0] | 10.0 [7.0 to 13.0] | 9.0 [6.0 to 13.0]
Hypertension [Count of Participants; unit: Participants] | 80 | 38 | 118
Heart failure [Count of Participants; unit: Participants] | 17 | 7 | 24
History of myocardial infarction [Count of Participants; unit: Participants] | 15 | 6 | 21
Chronic obstructive pulmonary disorder [Count of Participants; unit: Participants] | 15 | 7 | 22
Asthma [Count of Participants; unit: Participants] | 15 | 7 | 22
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 7 | 0 | 7
  Former smoker | 46 | 26 | 72
  Lifelong nonsmoker | 99 | 48 | 147
  Unknown | 9 | 8 | 17
Diabetes [Count of Participants; unit: Participants] | 45 | 30 | 75
History of cancer [Count of Participants; unit: Participants] | 22 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Ventilation or Death
Description: Time from administration of the investigational agent (or placebo) to requiring mechanical ventilation and intubation, or death for subjects who die prior to intubation. The percentages of patients who have been intubated or died as of day 14 and day 28 are estimated from the Kaplan-Meier curve.
Time Frame: 28 days
Population: Modified intention-to-treat (mITT) population, which includes 242 patients (161 in the tocilizumab group and 81 in the placebo group) who underwent randomization and received either tocilizumab or placebo before intubation or death
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 161 | 81
percentage of patients with event
  14 days | 9.9 [6.2 to 15.7] | 10.0 [5.1 to 18.9]
  28 days | 10.6 [6.7 to 16.6] | 12.5 [6.9 to 22.0]
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.64, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.38 to 1.81]

2. Secondary Outcome: Clinical Worsening on Ordinal Scale
Description: Time from administration of the investigational medication (or placebo) to at least one point worsening on the clinical improvement scale for subjects requiring supplemental oxygen (score >= 3) at baseline, or at least two point worsening otherwise (score = 2 at baseline). The percentages of patients who have worsened as of day 14 and day 28 are estimated from the Kaplan-Meier curve.
  Ordinal Scale
  1. Discharged
  2. Non-ICU hospital ward not requiring supplemental oxygen
  3. Non-ICU hospital ward requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring ECMO or mechanical ventilation and additional organ support
  7. Death
Time Frame: 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 161 | 81
percentage of patients with event
  Day 14 | 18.0 [12.9 to 24.9] | 14.9 [8.7 to 24.7]
  Day 28 | 19.3 [14.0 to 26.2] | 17.4 [10.7 to 27.7]
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.73, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.59 to 2.10]

3. Secondary Outcome: Discontinuation of Supplemental Oxygen Among Patients Receiving it at Baseline
Description: Time from administration of the investigational agent (or placebo) to absence of the need for supplemental oxygen among those who require at least supplemental oxygen at baseline. The percentages of patients who have discontinued supplemental oxygen as of day 14 and day 28 are estimated from the Kaplan-Meier curve.
Time Frame: 28 days
Population: A subset of 204 patients from the modified intention-to-treat (mITT) population who required at least supplemental oxygen at baseline. 138 patients in the tocilizumab group and 66 patients in the placebo group required at least supplemental oxygen at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 138 | 66
percentage of patients with event
  Day 14 | 75.4 [67.9 to 82.2] | 78.8 [68.3 to 87.7]
  Day 28 | 82.6 [75.9 to 88.4] | 84.9 [75.2 to 92.2]
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.69, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.67 to 1.30]

4. Other Pre Specified Outcome: Duration of Supplemental Oxygen
Description: Time from initiation of supplemental oxygen to end of supplemental oxygen use during 28-day study follow-up period. We includes all subjects in the analysis by assigning all subjects who did not receive supplemental oxygen a value of 0. Subjects who died prior to discontinuation of supplemental oxygen were given a value of the number of days from when supplemental oxygen began until the end of the follow-up period.
Time Frame: 28 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 161 | 81
days | 4.0 [1.8 to 11.6] | 3.9 [1.1 to 9.2]

5. Other Pre Specified Outcome: Duration of Mechanical Ventilation
Description: Time from initiation of mechanical ventilation to end of mechanical ventilation during 28-day study follow-up period, among patients who received mechanical ventilation. Event times of patients who died without discontinuation of mechanical ventilation were censored at 28 days. Median and inter-quartile range (IQR) were estimated using Kaplan-Meier curves. The upper limit for the IQR was not reached for both arms and entered as 28 in the outcome measure data table.
Time Frame: 28 days
Population: A subset of 19 patients from the modified intention-to-treat (mITT) population who received mechanical ventilation during the study follow-up period. 11 patients in the tocilizumab group and 8 patients in the placebo group received mechanical ventilation.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 11 | 8
days | 15.0 [12.6 to NA] — The upper limit for the IQR was not reached in the tocilizumab group. | 27.9 [16.3 to NA] — The upper limit for the IQR was not reached in the placebo group.

6. Other Pre Specified Outcome: Mortality
Description: Time from administration of the investigational agent (or placebo) to death. The percentage of patients who have died as of day 14 and day 28 are estimated from the Kaplan-Meier curve.
Time Frame: 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 161 | 81
percentage of patients with event
  Day 14 | 4.4 [2.1 to 8.9] | 1.3 [0.2 to 8.7]
  Day 28 | 5.6 [3.0 to 10.5] | 3.8 [1.2 to 11.3]

7. Other Pre Specified Outcome: ICU Admission or Death Among Those Not in the ICU at the Time of Administration of Investigational Agent (or Placebo)
Description: The percentage of subjects requiring ICU admission between baseline and 28 days is calculated by dividing the number of subjects requiring ICU admission over their hospitalization by the number of evaluable subjects (i.e., the number of subjects not in the ICU at the time of investigational treatment administration).
Time Frame: 28 days
Population: A subset of 233 patients from the modified intention-to-treat (mITT) population who were not in the ICU at baseline. 157 patients in the tocilizumab group and 76 patients in the placebo group were not in the ICU at baseline.
Measure: Number; unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 157 | 76
percentage of patients with event | 15.9 | 15.8

8. Other Pre Specified Outcome: Hospital Discharge
Description: Time from administration of the investigational medication (or placebo) to initial hospital discharge. Event times for patient who die are censored at day 29 to indicate that they never left the hospital during the follow-up period. The percentages of patients who were discharged as of day 14 and day 28 are estimated from the Kaplan-Meier curve.
Time Frame: 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 161 | 81
percentage of patients with event
  Day 14 | 86.3 [80.6 to 91.1] | 81.5 [72.4 to 89.0]
  Day 28 | 91.3 [86.3 to 95.0] | 88.9 [81.0 to 94.5]

9. Other Pre Specified Outcome: Clinical Improvement on Ordinal Scale
Description: Time to first improvement from administration of the investigational agent (or placebo) of at least 2 points (or the maximum amount) on the ordinal scale. Event times for patients who died prior to reaching this endpoint are censored at 29 days.
  Ordinal Scale
  1. Discharged
  2. Non-ICU hospital ward not requiring supplemental oxygen
  3. Non-ICU hospital ward requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring ECMO or mechanical ventilation and additional organ support
  7. Death
Time Frame: 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 161 | 81
percentage of patients with event
  Day 14 | 86.3 [80.6 to 91.1] | 81.5 [72.4 to 89.0]
  Day 28 | 91.3 [86.3 to 95.1] | 88.9 [81.0 to 94.5]

ADVERSE EVENTS:
Time Frame: 0-28 days. An AE is any unfavorable and unintended sign (including an abnormal laboratory finding),symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
Description: An SAE
  * death
  * It is life threatening
  * It requires or prolongs inpatient hospitalization.
  * It results in persistent or significant disability/incapacity
  * It results in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the IMP.
  * It is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the subject or may require medical/surgical intervention to prevent one of the outcomes listed above).
Arm/Group | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 9/161 | 4/82
Serious Adverse Events (participants affected / at risk) | 19/161 | 8/82
Other Adverse Events (participants affected / at risk) | 20/161 | 26/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=161) | Placebo (N=82)
Elevated liver function test: Alanine aminotransferase (Hepatobiliary disorders) | 1 (1) | 1 (1)
Elevated liver function test: Aspartate transaminase (Hepatobiliary disorders) | 1 (1) | 1 (1)
Arterial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Deep venous thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Infection (Infections and infestations) | 4 (4) | 6 (6)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Continued anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) — patient continues inpatient due to refusal of food and IV medications - prolong
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) — after standing up - BP 79/60. IV fluid bolus given with BP back to 120s again
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Elevated Partial Thromboplastin Time (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Low output from nephrostomy tube (Renal and urinary disorders) | 1 (1) | 0 (0) — decreased urine output from his right-sided nephrostomy tube
Patient re-hospitalized because dialysis could not be arranged any other way (Renal and urinary disorders) | 1 (1) | 0 (0)
Hip fracture requiring hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheostomy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — patient experienced episode of tachypnea post bed bath(Grade 3
Parasthesia (Nervous system disorders) | 0 (0) | 1 (1) — there was noted change in neurology exam with patient now not withdrawing to pain in upper extremity
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — resulting in PEG placement
respiratory failure and intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — to the 40's to the point of brief asystole
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypothermia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization for Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Grade 3: Rash/allergic reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=161) | Placebo (N=81)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — (including elevated creatinine, decreased GFR)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Decreased poly(ADP-ribosyl)ation (Immune system disorders) | 1 (1) | 0 (0)
decreased white blood cell count (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Increased alkaline phosphatase (Renal and urinary disorders) | 1 (1) | 1 (1)
Paroxysmal Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Pruritic Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Worsening confusion (Nervous system disorders) | 1 (1) | 1 (1)
worsening lower extremity wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
decreased hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
acute kidney injury with AGMA and hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
FALL WITH ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
hypomagnesemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mild edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Mucus plugging (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT04356937/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT04356937/SAP_001.pdf